CLINICAL TRIAL: NCT00348335
Title: Efficacy of Topical Cyclosporin 0.05% for the Treatment of Ocular Rosacea
Brief Title: Efficacy of Topical Cyclosporin for Ocular Rosacea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ophthalmic Consultants of Long Island (Other)
Collaborators: Allergan (Industry)
Responsible Party: Dr. Eric Donnenfeld, OCLI
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 32,133
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2011-07-29 (Estimated); Status verified 2011-07

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1: Restasis (Active Comparator)
  Interventions: Drug: Cyclosporine 0.05%
- 2: Refresh Endura (Active Comparator)
  Interventions: Drug: Ocular lubricant

INTERVENTIONS:
Drug: Cyclosporine 0.05%
  Arms: 1: Restasis
Drug: Ocular lubricant
  Arms: 2: Refresh Endura

SUMMARY:
The purpose of this study is to determine whether Restasis (topical cyclosporin) is effective in the treatment of ocular rosacea

DETAILED DESCRIPTION:
The study is designed to compare the efficacy of topical cyclosporin (Restasis) with that of Refresh Endura for the treatment of the signs and symptoms of ocular rosacea in patients presently controlled on topical corticosteroids

ELIGIBILITY:
Inclusion Criteria:

* Patient at least 18 years old, but younger than 65
* Diagnosis of acne rosacea
* Active ocular rosacea based on lid findings of meibomian gland dysfunction with lid telangiectasia and hyperemia of at least 2+
* Schirmers test of greater than 5mm in at least 1 eye
* If patient currently using lid hygiene must maintain regimen during study
* Stop oral antibiotics at least 4 weeks prior

Exclusion Criteria:

* Use of topical cyclosporin within last 90 days
* Visual acuity of 20/100 or better in both eyes
* Pregnant or lactating females
* Active ocular infection
* Scarring of central cornea
* Eyelid defects,abnormal lid positioning or lagophthalmos
* Flax seed or Fish oil supplements within last 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2006-06; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
hyperemia | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: John R Wittpenn, MD, Principal Investigator — Ophthalmic Consultants of Long Island
Locations (1):
- 2500 Rte 347 Bldg 24, Stony Brook, New York, United States